CLINICAL TRIAL: NCT06855368
Title: Brain Connectivity and Complexity Parameters to Monitor Disease Progression in Dementia Patients and Antiinflammatory Nanotherapeutics in a Preclinical Model of Alzheimer's Disease
Brief Title: Biomarkers for Monitoring Dementia Progression
Acronym: ADvance
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 22/25
Record Dates: First submitted 2025-01-29; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
Keywords: EEG; functional connectivity; neuroinflammation; nanoparticles
MeSH Terms: conditions — Alzheimer Disease; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AD
- MCI
- HC

SUMMARY:
The variable course of Alzheimer's disease (AD) and the paucity of adequate cures urges to implement new strategies for its early detection and clinical intervention. Studying the etiopathogenesis and pathophysiological mechanisms of AD is a necessary prerequisite for the development of new biomarkers and innovative therapies. Contrarily to anatomical structures, cortical connectivity networks are already deteriorated in early AD and could be a reliable marker of early cognitive decline. Our aim is to characterize the neurophysiological parameters in mild AD, in patients with mild cognitive impairment and in matched healthy subjects to identify discriminating criteria. Concurrently, the study of AD onset and progression in a mouse model, will allow evaluating the causal effect of inflammation on disease progression and to develop a new class of biomimetic anti-inflammatory nanoparticles formulated to have the intrinsic ability to induce brain's activated microglia to an M2 phenotype.

ELIGIBILITY:
Inclusion Criteria:

* mild AD and patients with mild cognitive impairment (MCI).

Exclusion Criteria:

* major psychosis, genetic, metabolic and other neurological disorders, acute or chronic non-compensated medical illness
* any medical or drug-related condition affecting cognitive or mood status
* history or current alcohol/illicit drug abuse.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 AD and 100 MCI individuals from the dementia clinical centres of North Sardinia and local sections of patients¿ associations and 100 HC will be recruited for the study. To investigate past/present health status and medications, baseline medical screening will be performed by general clinical and anthropometric examinations
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-05-17 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Disease-Associated Phenotypes in MCI and AD | through study completion, an average of 1 year
Identification of Disease-Associated Early Interventions in MCI and AD | through study completion, an average of 1 year
Predictive Power of EEG-Based Brain Network Analyses for MCI to AD Conversion | through study completion, an average of 1 year
  EEG power spectral density
Evaluation of Targeting Efficiency of Activated vs Native Leukosomes in Brain Inflammation | through study completion, an average of 1 year
Evaluation Trafficking Kinetics of Activated vs Native Leukosomes in Brain Inflammation | through study completion, an average of 1 year
Assessment of Activated Leukosomes in Inducing Anti-Inflammatory Polarization of Macrophages | through study completion, an average of 1 year
Assessment of Activated Leukosomes in Glial Cells | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS San Raffaele, Roma
  - Azienda Ospedaliero-Universitaria di Sassari, Sassari